CLINICAL TRIAL: NCT02503774
Title: A Phase 1 Multicenter, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI9447 Alone and in Combination With MEDI4736 in Adult Subjects With Select Advanced Solid Tumors
Brief Title: MEDI9447 Alone and in Combination With MEDI4736 in Adult Participants With Select Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6070C00001
Record Dates: First submitted 2015-07-06; First posted 2015-07-21 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Solid Tumors
Keywords: Solid Tumors,; MEDI9447,; oleclumab,; MEDI4736,; durvalumab,; CD73,; programmed death ligand-1 (PD-L1),; epidermal growth factor receptor mutant (EGFRm) non-small cell lung cancer (NSCLC),; immunotherapy,; pancreatic,; colorectal
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Dose-escalation: Oleclumab Dose 1 (Experimental): Participants will receive oleclumab Dose 1 intravenously (IV) every two weeks (Q2W) until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab
- Dose-escalation: Oleclumab Dose 2 (Experimental): Participants will receive oleclumab Dose 2 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab
- Dose-escalation: Oleclumab Dose 3 (Experimental): Participants will receive oleclumab Dose 3 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab
- Dose-escalation: Oleclumab Dose 4 (Experimental): Participants will receive oleclumab Dose 4 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab
- Dose-escalation: Oleclumab Dose 1 + Durvalumab Dose 1 (Experimental): Participants will receive oleclumab Dose 1 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-escalation: Oleclumab Dose 2 + Durvalumab Dose 1 (Experimental): Participants will receive oleclumab Dose 2 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-escalation: OleclumabDose 3 + Durvalumab Dose 1 (Experimental): Participants will receive oleclumab Dose 3 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-escalation: OleclumabDose 4 + Durvalumab Dose 1 (Experimental): Participants will receive oleclumab Dose 4 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-expansion (CRC): Oleclumab Dose 4 + Durvalumab Dose 1 (Experimental): Participants with previously treated microsatellite stable-colorectal cancer (MSS-CRC) will receive oleclumab Dose 4 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-expansion (Pancreatic adenocarcinoma): Oleclumab Dose 4+ Durvalumab Dose 1 (Experimental): Participants with previously treated pancreatic adenocarcinoma will receive oleclumab Dose 4 IV Q2W followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab
- Dose-expansion (NSCLC): Oleclumab Dose 4 + Durvalumab Dose 1 (Experimental): Participants with previously treated EGFRm NSCLC will receive oleclumab Dose 4 IV followed by durvalumab Dose 1 IV Q2W until confirmed disease progression, unacceptable toxicity, withdrawal of consent, or development of other reason for treatment discontinuation, whichever occurs first.
  Interventions: Drug: Oleclumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Oleclumab — Participants will receive IV infusion of oleclumab as stated in arms' description.
Drug: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arms' description.
  Arms: Dose-escalation: Oleclumab Dose 1 + Durvalumab Dose 1; Dose-escalation: Oleclumab Dose 2 + Durvalumab Dose 1; Dose-escalation: OleclumabDose 3 + Durvalumab Dose 1; Dose-escalation: OleclumabDose 4 + Durvalumab Dose 1; Dose-expansion (CRC): Oleclumab Dose 4 + Durvalumab Dose 1; Dose-expansion (NSCLC): Oleclumab Dose 4 + Durvalumab Dose 1; Dose-expansion (Pancreatic adenocarcinoma): Oleclumab Dose 4+ Durvalumab Dose 1

SUMMARY:
The purpose of this study is to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of MEDI9447 Alone and in Combination with MEDI4736 in Adult Participants with Select Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Adult participants; age ≥ 18
* Written and signed informed consent must be obtained
* Have histologic or cytologic documentation of solid tumor including EGFRm NSCLC
* Participants must have at least 1 lesion that is measurable using RECIST guidelines
* Participants must consent to provide archived tumor specimens or tumor biopsies for correlative biomarker studies.
* Eastern Cooperative Oncology Group performance score of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Prior treatment with tumor necrosis factor receptor superfamily agonists including OX40, CD27, CD137 (4-1BB), CD357 (GITR). One cohort also excludes anti CTLA-4, PD-L1, and anti PD-L1.
* Participants who have received prior therapy with regimens containing CTLA-4, PD-L1, or PD-1 antagonists may be permitted to enroll under certain conditions
* Cardiac or peripheral vascular disease meeting any of the following criteria:

  * Past history of myocardial infarction in the prior 12 months
  * Past history of stroke or transient ischemic attack requiring medical therapy
  * Congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification
* Grade 3 or greater edema (eg, peripheral, pulmonary)
* History of Grade 3 or greater thromboembolic events in the prior 12 months
* Participants with active tuberculosis are ineligible. In settings where there is clinical or radiographic evidence of tuberculosis, active disease must be ruled out
* Active or prior documented autoimmune or inflammatory disorders
* Untreated central nervous system (CNS) metastatic disease
* Known positive for human immunodeficiency virus (HIV), chronic or active hepatitis B or active hepatitis A or C
* Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast that has been surgically cured
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active peptic ulcer disease or gastritis, uncontrolled hypertension, uncontrolled diabetes, or psychiatric illness/social situations that would limit compliance with study requirement

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) in Dose-escalation Phase | From Day 1 to Day 28 after first dose of study drug
  A DLT was defined as any Grade 3 or higher treatment-related toxicity that occurred during the DLT-evaluation period, which included any Grade 4 immune-mediated adverse event (imAE), any >= Grade 3 colitis, any Grade 3 or 4 non-infectious pneumonitis irrespective of duration, any Grade 3 imAE (excluding colitis or pneumonitis, did not downgrade to <= Grade 2 within 3 days after onset of the event despite maximal medical supportive care including systemic corticosteroids or did not downgrade to <= Grade 1 or baseline within 14 days), liver transaminase elevation >= 5 × but <= 8 × upper limit of normal (ULN) that did not downgrade to Grade 2 within 5 days after onset with optimal medical management (including systemic corticosteroids), transaminase elevation > 8 × ULN or total bilirubin (TBL) > 5 × ULN regardless of duration or reversibility, or any increase in aspartate aminotransferase or alanine aminotransferase > 3 × ULN and concurrent increase in TBL > 2 × ULN (Hy's Law).
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | From Day 1 through 200.1 weeks (corresponding to maximum observed duration)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs | From Day 1 through 200.1 weeks (corresponding to maximum observed duration)
  Participants with abnormal laboratory parameters reported as TEAEs are reported. Laboratory analysis included hematology, clinical chemistry, thyroid function tests, coagulation, and urinalysis.
Number of Participants With Abnormal Vital Signs Reported as TEAEs | From Day 1 through 188.1 weeks (corresponding to maximum observed duration)
  Participants with abnormal vital signs (temperature, blood pressure, pulse rate, and respiratory rate) reported as TEAEs are reported.
Number of Participants With Change From Baseline in QTcF | Baseline (prior to Day 1 dose) through 188.1 weeks (corresponding to maximum observed duration)
  Number of participants with change from Baseline in QTcF (> 60 msec and > 90 msec) is reported.

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response (OR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 | Baseline (Days -28 to -1) through 53 months (corresponding to maximum observed duration)
  The OR is defined as confirmed complete response (CR) or confirmed partial response (PR) based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and the non-target lesion at least stable with no evidence of new lesions. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression in-between. Percentage of participants with OR are reported.
Percentage pf Participants With Disease Control (DC) per RECIST v1.1 | Baseline (Days -28 to -1) through 53 months (corresponding to maximum observed duration)
  The DC is defined as CR, PR, or stable disease (SD) which was maintained by >= 8 weeks from the start of treatment. The SD is defined as neither sufficient shrinkage of target lesion to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum of diameters while on study and non-progressive disease and not evaluable or no non-target lesion. The CR is defined as disappearance of all target and non-target lesions, and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and the non-target lesion at least stable with no evidence of new lesions. Percentage of participants with DC at >= 8 weeks, >= 16 weeks, and >= 24 weeks are reported.
Duration of Response (DoR) per RECIST v1.1 | Baseline (Days -28 to -1) through 53 months (corresponding to maximum observed duration)
  The DoR is defined as the duration from the first documentation of OR (confirmed CR or PR) to the first documented PD or death due to any cause, whichever occurred first. The CR is defined as disappearance of all target and non-target lesions, and no new lesions. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline, and the non-target lesion at least stable with no evidence of new lesions. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression or not evaluable response in-between. The PD is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The DoR was estimated using Kaplan-Meier method.
Progression-Free Survival (PFS) | Baseline (Days -28 to -1) through 53 months (corresponding to maximum observed duration)
  The PFS is defined as the time from the start of study treatment until the documentation of PD based on RECIST version 1.1 or death due to any cause, whichever occurred first. The PD is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. The PFS was estimated using Kaplan-Meier method.
Overall Survival (OS) | Baseline (Days -28 to -1) through 53 months (corresponding to maximum observed duration)
  The OS is defined as the time from the start of treatment with study drug until death due to any cause. The OS was estimated using Kaplan-Meier method.
Maximum Observed Serum Concentration (Cmax) of MEDI9447 | Day 1 (pre-dose, and 10 minutes and 2 hours post end of infusion), Day 57 (pre-dose and 10 minutes post end of infusion)
  The Cmax of MEDI9447 (oleclumab) for Cycle 1 and at steady state (Day 57) are reported.
Area Under the Serum Concentration Time Curve From 0 To 14 Days Post First Dose [AUC(0-14)] of MEDI9447 | Day 1 (pre-dose; 10 minutes and 2 hours post end of infusion)
  The AUC(0-14) of MEDI9447 is reported.
Time To Maximum Observed Serum Concentration (Tmax) of MEDI9447 | Day 1 (pre-dose; 10 minutes, 2 hours post end of infusion); Day 57 (pre-dose; 10 minutes post end of infusion)
  The Tmax of MEDI9447 for Cycle 1 and at steady state (Day 57) of MEDI9447 are reported.
Observed Lowest Serum Concentration Reached Before the Next Dose (Ctrough) of MEDI9447 | Day 1 (pre-dose; 10 minutes, 2 hours post end of infusion); Day 57 (pre-dose; 10 minutes post end of infusion)
  The Ctrough of MEDI9447 for Cycle 1 and at steady state (Day 57) of MEDI9447 are reported.
Accumulation Ratio for Cmax (Rac Cmax) of MEDI9447 | Day 57 (pre-dose; 10 minutes post end of infusion)
  The Rac Cmax of MEDI9447 for Cycle 1 and at steady state (Day 57) of MEDI9447 is reported.
Accumulation Ratio for Ctrough (Rac Ctrough) of MEDI9447 | Day 57 (pre-dose; 10 minutes post end of infusion)
  The Rac Ctrough of MEDI9447 is reported.
Cmax of MEDI4736 | Day 1 (prior to start of MEDI9447 infusion and 10 minutes post end of MEDI4736 infusion)
  The Cmax of MEDI4736 (durvalumab) is reported.
Tmax of MEDI4736 | Day 1 (prior to start of MEDI9447 infusion and 10 minutes post end of MEDI4736 infusion)
  The Tmax of MEDI4736 is reported.
Ctrough of MEDI4736 | Day 1 (prior to start of MEDI9447 infusion and 10 minutes post end of MEDI4736 infusion), Day 57 (prior to start of MEDI9447 infusion)
  The Ctrough of MEDI4736 for Cycle 1 and at steady state (Day 57) are reported.
Rac Ctrough of MEDI4736 | Day 57 (prior to start of MEDI4736 infusion)
  The Rac Ctrough of MEDI4736 is reported.
Number of Participants With Positive Anti-Drug Antibody Response (ADA) to MEDI9447 | Day 1 through 192.3 weeks (Days 1 , 29, and 57, EOT, and 30 days post end of treatment)
  Number of participants with positive ADA to MEDI9447 is reported. Persistent positive was defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive was defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with < 16 weeks between first and last positive).
Number of Participants With Positive ADA to MEDI4736 | Day 1 through 200.1 weeks (Day 1 through 192.3 weeks (Days 1 , 29, and 57, EOT, and 30 days post end of treatment)
  Number of participants with positive ADA to MEDI4736 is reported. Persistent positive was defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive was defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with < 16 weeks between first and last positive).

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (16):
- United States (11):
  - Research Site, La Jolla, California
  - Research Site, New Haven, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, St Louis, Missouri
  - Research Site, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
- Australia (4):
  - Research Site, Camperdown
  - Research Site, Parkville
  - Research Site, St Leonards
  - Research Site, Woolloongabba
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Bendell J, LoRusso P, Overman M, Noonan AM, Kim DW, Strickler JH, Kim SW, Clarke S, George TJ, Grimison PS, Barve M, Amin M, Desai J, Wise-Draper T, Eck S, Jiang Y, Khan AA, Wu Y, Martin P, Cooper ZA, Elgeioushi N, Mueller N, Kumar R, Patel SP. First-in-human study of oleclumab, a potent, selective anti-CD73 monoclonal antibody, alone or in combination with durvalumab in patients with advanced solid tumors. Cancer Immunol Immunother. 2023 Jul;72(7):2443-2458. doi: 10.1007/s00262-023-03430-6. Epub 2023 Apr 5. PMID 37016126
- [Derived] Hay CM, Sult E, Huang Q, Mulgrew K, Fuhrmann SR, McGlinchey KA, Hammond SA, Rothstein R, Rios-Doria J, Poon E, Holoweckyj N, Durham NM, Leow CC, Diedrich G, Damschroder M, Herbst R, Hollingsworth RE, Sachsenmeier KF. Targeting CD73 in the tumor microenvironment with MEDI9447. Oncoimmunology. 2016 Jul 11;5(8):e1208875. doi: 10.1080/2162402X.2016.1208875. eCollection 2016 Aug. PMID 27622077
- See also: study-synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6070C00001&attachmentIdentifier=87228817-1164-4242-9e13-7f33fe991dd0&fileName=D6070C00001-study-synopsis_Redacted_KH.pdf&versionIdentifier=